CLINICAL TRIAL: NCT06373731
Title: ReNEW: A Phase 3, Double-Masked, Placebo-Controlled Clinical Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of Subcutaneous Injections of Elamipretide in Subjects Who Have Dry Age-Related Macular Degeneration (Dry AMD)
Brief Title: ReNEW:Phase 3 Study of Efficacy, Safety & Pharmacokinetics of Subcutaneous Injections of Elamipretide in Subjects With Dry Age-Related Macular Degeneration (Dry AMD)
Acronym: ReNEW
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIAM-301
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Age Related Macular Degeneration (ARMD)
Keywords: dAMD, Dry AMD, dryAMD; Macular degeneration; non-central geographic atrophy, GA; MTP-131; elamipretide; Non- Intravitreal, Non- gene therapy
MeSH Terms: conditions — Macular Degeneration | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized (2:1) to once daily 40 mg SC of elamipretide or placebo for 96 weeks of treatment by a central randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial personnel and subjects will be masked to treatment until the database is locked at the end of the trial, unless noted below. The Investigator will contact the Sponsor Medical Monitor prior to unmasking any subject's treatment sequence unless in the instance of a medical emergency. In case of an immediate medical emergency, or if directed by the Sponsor, and only if the information is required by the Investigator to manage a subject's AE, a subject's treatment assignment may be unmasked prematurely using the computerized system. The Sponsor must be notified as soon as possible regarding the reason for unmasking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elamipretide (Experimental): Subjects will receive once daily subcutaneous doses of 40mg elamipretide for 96 weeks
  Interventions: Drug: Elamipretide
- Placebo (Placebo Comparator): Subjects will receive once daily subcutaneous doses of placebo for 96 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elamipretide — Subjects will receive once daily SC doses of 40 mg elamipretide for 96 weeks
  Other Names: Elamipretide HCL
  Arms: Elamipretide
Drug: Placebo — Subjects will receive once daily SC doses of Placebo 96 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy, safety and pharmacokinetics of elamipretide in subjects with dry age-related macular degeneration (AMD). The main questions it aims to answer are: what is the rate of change in the macular area of photoreceptor loss in subjects who receive a daily dose of elamipretide compared with those who receive a look-alike substance that contains no active drug, and what is the safety and tolerability of elamipretide daily subcutaneous injections. Participants will receive either once daily subcutaneous doses of 40mg elamipretide or placebo and the two treatment groups will be compared.

DETAILED DESCRIPTION:
The ReNEW (SPIAM-301) trial is a phase 3, randomized, double-masked, parallel-group, placebo-controlled clinical trial to evaluate the efficacy, safety, and pharmacokinetics of a once daily subcutaneous (SC) injection of elamipretide in subjects who have dry AMD. Subjects will be randomized (2:1) to once daily SC doses of 40 mg elamipretide, or placebo for 96 weeks of treatment by a central randomization and stratified by SD-OCT device type (Heidelberg SPECTRALIS®, ZEISS CIRRUS®) and baseline macular area of photoreceptor loss, defined as an ellipsoid zone-retinal pigment epithelium (EZ-RPE) thickness of 0μm assessed by SD-OCT and ellipsoid zone (EZ) mapping (High Strata ≥ 5.1mm2, Low Strata <5.1mm2).

Primary Objective

* Evaluate the efficacy of once daily subcutaneous (SC) injections of elamipretide in subjects who have dry age-related macular degeneration (AMD) Secondary Objectives
* Evaluate the safety and tolerability of once daily SC injections of elamipretide
* Evaluate the Pharmacokinetic (PK) profile of elamipretide and its metabolites

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all the inclusion criteria at the Screening and Baseline Visit (unless otherwise specified) to be eligible for inclusion in the trial.

1. Adults ≥ 55 years of age with at least 1 eye with dry AMD with photoreceptor loss, as determined at the Screening Visit by the presence of extrafoveal geographic atrophy (GA), as determined by the Reading Center primarily by fundus autofluorescence (FAF). For this trial, extrafoveal GA is defined as:

   1. well-demarcated area(s) of GA
   2. All GA lesions must be at least 150 μm from foveal center Note: The fellow eye may have any of the following: no AMD, AMD without GA, AMD with GA, CNV AMD, or foveal GA (ongoing treatment with anti-angiogenic therapies and/or complement inhibitor therapies in the fellow eye is allowable)

   Ocular conditions - Study Eye:
2. GA in the study eye at the Screening Visit may be multi-focal, but the cumulative GA lesion and size (by FAF, as determined by the Reading Center) must:

   1. be ≥ 0.50 mm2 and ≤ 10.16 mm2 AND
   2. reside completely within the FAF 30- or 35-degree image
3. BCVA by Early Treatment Diabetic Retinopathy Study (ETDRS) score of ≥ 55 letters in the study eye
4. LL BCVA by ETDRS score of ≥ 10 letters in the study eye
5. LLD (defined as the difference between BCVA and LL BCVA) of > 5 letters in the study eye
6. Sufficiently clear ocular media, adequate pupillary dilation, fixation to permit quality fundus imaging, and ability to cooperate sufficiently for adequate ophthalmic visual function testing and anatomic assessment in the study eye

   Systemic and General Criteria:
7. Able to administer IMP or have an appropriate designee who can administer the IMP (i.e., a capable family member or a caregiver)
8. Able to provide informed consent and willing to comply with all site visits, examinations, daily IMP administrations and dosing diary entries, and other conditions of the trial protocol
9. Women of childbearing potential must agree to use 1 of the following methods of contraception from the date they sign the ICF until 28 days after the last dose of IMP:

   1. Abstinence, when it is in line with the preferred and usual lifestyle of the subject; Subject agrees to use a highly effective method of contraception should they become sexually active
   2. Relationships with male partners who have been surgically sterilized by vasectomy (the vasectomy procedure must have been conducted at least 60 days prior to the Screening Visit)
   3. Barrier method (e.g., condom or occlusive cap) with spermicidal foam/gel/film/cream AND either hormonal contraception (oral, implanted, or injectable) or an intrauterine device or system Note: Non-childbearing potential is defined as surgical sterilization (e.g., bilateral oophorectomy, hysterectomy, or tubal ligation) or postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to the Screening Visit).
10. Male subjects with female partners of childbearing potential must be willing to use a highly effective method of contraception (e.g., abstinence, dual method of contraception) from the date they sign the ICF until 28 days after the last dose of IMP

Exclusion Criteria:

Subjects who meet any of the following criteria at the Screening and Baseline Visit (unless otherwise specified) will be excluded from the trial:

Ocular Conditions - Study Eye:

1. The absence of observable hyper-FAF at the margins of the GA in the study eye at the Screening Visit by the Reading Center
2. Atrophic retinal disease of causality other than AMD including myopia-related maculopathy and monogenetic macular dystrophies including pattern dystrophy and adult-onset Stargardt disease in the study eye
3. Evidence of exudative AMD or CNV in the study eye by history or FA , as determined by the Reading Center
4. Presence of retinal vein occlusion in the study eye
5. Presence of vitreous hemorrhage in the study eye
6. History of retinal detachment in the study eye
7. History of macular hole (stages 2 to 4) in the study eye
8. Presence of an epiretinal membrane and/or vitreomacular traction in the study eye that causes distortion of the retinal contour
9. Presence of any retinal pathology in the study eye that prohibits outer retinal quantification and EZ mapping, as determined at the Screening Visit by the Reading Center
10. At the Screening Visit, advanced glaucoma resulting in a cup to disc ratio of > 0.8 in the study eye
11. History of glaucoma filtration surgery or uncontrolled glaucoma at Baseline Visit in the opinion of the Investigator OR currently using ≥ 3 medications (Minimally invasive glaucoma surgeries (e.g., MIGS) are allowable) Note: Combination medications count as 2 medications.
12. Presence of visually significant cataract OR presence of significant posterior capsular opacity in the setting of pseudophakia Note: Significant cataract is defined as ≥ +3 nuclear sclerosis based upon the scale below or any Posterior Subcapsular Cataract in the study eye. The Sponsor, or its designee, will supply the clinical trial sites with a copy of the standard photographs. Grade Description

    * 1 Opacity is absent
    * 2 Opacity is present, but less than Nuclear Standard Photograph #2
    * 3 Opacity is present, and as severe as or worse than Nuclear Standard Photograph #2 Source: (Chew 2010)
13. Presence of significant keratopathy or any other media or corneal opacity that would cause scattering of light or alter visual function, especially in LL conditions in the study eye
14. Ocular incisional or laser surgery (including cataract surgery) in the study eye within 90 days before the Baseline Visit
15. YAG laser capsulotomy in the study eye within 30 days before the Baseline Visit
16. Aphakia in the study eye
17. History of vitrectomy surgery, submacular surgery, or any vitreoretinal surgery in the study eye
18. Prior treatment with Visudyne® (verteporfin) ocular photodynamic therapy, external-beam radiation therapy (for intraocular conditions), or transpupillary thermotherapy in the study eye
19. History of subthreshold laser treatment or other forms of photobiomodulation for AMD in the study eye
20. Intravitreal drug delivery in the past 60 days or 5-half-lives from the Baseline Visit of the injected drug whichever is longer (e.g., intravitreal corticosteroid injection, anti-angiogenic drugs, or device implantation) in the study eye
21. Intravitreal drug delivery of a complement inhibitor in the past 6 months from the Baseline Visit in the study eye
22. Concurrent disease in the study eye that could require medical or surgical intervention during the trial

    Ocular conditions - Either Eye:
23. Presence or a history of diabetic retinopathy in either eye (a history of diabetes mellitus without retinopathy is not a criterion for exclusion)
24. History of herpetic infection in either eye
25. Active uveitis and/or vitritis (grade trace or above) in either eye
26. History of idiopathic or autoimmune-associated uveitis in either eye
27. Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye

    Systemic Conditions:
28. Has a history of a systemic eosinophilic illness and/or an eosinophil count >1,000 cells x106/L (equivalent to >1 cell x 103/μL) at the Screening Visit
29. History of solid organ transplant
30. Any disease or medical condition that in the opinion of the Investigator would prevent the subject from successfully participating in the trial or might confound trial results
31. Current use of medications known to be toxic to the lens, retina, or optic nerve (e.g., deferoxamine, chloroquine/hydroxychloroquine [Plaquenil®], tamoxifen, phenothiazines, ethambutol, digoxin, and aminoglycosides)
32. eGFR of < 30 mL/min at the Screening Visit (using the CKD-EPI 2021 formula)

    General Conditions:
33. Participation in other investigational drug or device clinical trials within 30 days or 5 half-lives (whichever is longer) of Screening; or is currently enrolled in a non-interventional clinical trial that, in the opinion of the Investigator, may be potentially confounding to the results of the current trial
34. Women who are pregnant, planning to become pregnant, or breastfeeding/lactating
35. History of allergy to fluorescein that is not amenable to treatment
36. Inability to comply with trial or follow-up procedures
37. Inability to obtain CFP, FAF, and FA of sufficient quality to be analyzed and interpreted
38. Active malignancy or any other cancer from which the subject has been cancer-free for < 2 years. Localized squamous or non-invasive basal cell skin carcinomas are allowed, if appropriately treated prior to screening
39. History of allergic reaction to the investigational drug or any of its components
40. Prior participation in any elamipretide trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Week 48 Rate of change in the macular area of photoreceptor loss | Baseline, Week 48
  Rate of change in the macular area of photoreceptor loss (defined as an EZ-RPE thickness of 0μm) assessed by SD-OCT and EZ mapping at Week 48

SECONDARY OUTCOMES:
Week 72 Rate of change in the Macular area of photoreceptor loss | Baseline, Week 72
  Rate of change in the macular area of photoreceptor loss (defined as an EZ-RPE thickness of 0μm) assessed by SD-OCT and EZ mapping at Week 72
Week 96 Rate of change in the Macular area of photoreceptor loss | Baseline, Week 96
  Rate of change in the macular area of photoreceptor loss (defined as an EZ-RPE thickness of 0μm) assessed by SD-OCT and EZ mapping
Proportion of subjects gaining ≥ 10 letters (2 lines) in Low Luminance Best-Corrected Visual Acuity (LL BCVA) | Baseline, Week 48
  Proportion of subjects gaining ≥ 10 letters (2 lines) in Low Luminance Best- Corrected Visual Acuity (LL BCVA) from baseline at Week 48
Proportion of subjects gaining ≥ 15 letters in Low Luminance Best-Corrected Visual Acuity (LL BCVA) | Baseline, Week 48
  Proportion of subjects gaining ≥ 15 letters (3 lines) in LL BCVA from baseline at Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sathyanarayana, Study Director — Stealth BioTherapeutics
Locations (53):
- United States (31):
  - Associated Retina Consultants, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Sun City, Arizona
  - Retina Associates of Southern California, Huntington Beach, California
  - Retina Consultants of San Diego, Poway, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Orange County Retinal Medical Group, Santa Ana, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Connecticut Eye Consultants, P.C., Danbury, Connecticut
  - Vitreo Retinal Associates, Gainesville, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Associated Vitreoretinal and Uveitis Consultants, Carmel, Indiana
  - Mid Atlantic Retina Specialist, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Kellogg Eye Center, Ann Arbor, Michigan
  - Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - Retina Vitreous Center, Edmond, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Valley Retina Institute, McAllen, Texas
  - Texas Retina Associates of Plano, Plano, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Pacific Northwest Retina, PLLC, Silverdale, Washington
- Axon Clinical, s.r.o., Prague, Czechia
- Germany (3):
  - Augenzentrum am St. Franziskus-Hospital, Münster
  - Klinik und Poliklinik für Augenheilkunde- Universitätsklinik Regensburg, Regensburg
  - Department für Augenheilkunde, Tübingen
- Hungary (3):
  - University Of Debrecen Eye Center, Debrecen
  - Ganglion Medical Center, Pécs
  - University of Szeged, Department of Ophthalmology, Szeged
- Italy (5):
  - Hospital Luigi Sacco Ophthalmology Dept, Milan
  - IRRCS Ospendale San Raffaele, Milan
  - Policlinico Milano, Milan
  - Fondazione Policlinico Gemelli, Roma
  - Department of Ophthalmology, Azienda SanitariaUniversitaria Friuli Centrale, Udine
- New Zealand (2):
  - Southern Eye Specialists, Christchurch
  - Capital Eye Specialists, Wellington
- Spain (4):
  - Centro de Oftalmologia Barraquer, Barcelona
  - OMIQ Research, Barcelona
  - Fundacion Aiken de la Comunitat Valenciana, Valencia
  - Oftalvist, Valencia
- United Kingdom (4):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Eye Hospital, Bristol
  - University Hospitals of Leicester, Leicester Royal Infirmary, Leicester
  - Macular Services, Central Middlesex Hospital, NHS Foundation Trust, London
  - South Tyneside and Sunderland NHS Foundation Trust - Sunderland Eye Infirmary, Sunderland